CLINICAL TRIAL: NCT03603483
Title: Short Term Outcome of Aortic Root Enlargement in Management of Small Aortic Annulus Among Patients With Severe Valvular Aortic Stenosis
Brief Title: Aortic Root Enlargement in Aortic Valve Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed mahmoud ahmed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aortic root enlargement
Record Dates: First submitted 2018-03-08; First posted 2018-07-27 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Aortic Valve Replacement
Keywords: patients- prosthesis mismatching
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Aortic Root Enlargement in Patients with aortic stenosis with Small Aortic Annulus
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with sever aortic stenosis 1 (Active Comparator): Procedure: the patients will undergo aortic valve replacement with aortic root enlargement.
  Interventions: Procedure: procedure
- Patients with sever aortic stenosis 2 (Active Comparator): Procedure: the patients will undergo conventional aortic valve replacement
  Interventions: Procedure: procedure

INTERVENTIONS:
Procedure: procedure — Patients of sever aortic stenosis 1: increase the diameter of aortic anulus by prosthetic patch or pericardial patch.
  Patients of sever aortic stenosis 1:only conventional aortic valve prosthesis will be used

SUMMARY:
Aortic valve disease is a progressive illness that varies from minor valve thickening lacking obstruction of blood stream to severe calcification and alteration of the valve leading to weakened leaflet motion. Aortic valve replacement is a usual operation but can be complicated by a small aortic annulus requiring the insertion of an aortic valve prosthesis. Prosthesis-patient discrepancy results in worse outcomes.

DETAILED DESCRIPTION:
Prosthesis-patient discrepancy results in worse outcomes, including elevated left ventricular work, decreased left ventricular mass regression, and has also been linked with high mortality. Therefore, Aortic root posterior enlargement by autologous fixed pericardium to insert an Aortic valve prosthesis with size suitable to patient body surface area to avoid the previous worse outcome of patient prosthesis mismatch. In this study the investigators will try to identify the benefits of Aortic Root Enlargement in management of Small Aortic Annulus in Patients with severe valvular aortic stenosis

ELIGIBILITY:
Inclusion Criteria:

* 17-75 years old
* patients with sever aortic valve stenosis undergoing valve replacement surgery
* informed consent has been obtained

Exclusion Criteria:

* Planned off-pump cardiac surgery
* Patients required intra-aortic balloon pump
* under 17 years of age

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-15 (Estimated); Primary Completion 2019-03-28 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
Transthoracic echocardiographic measurement of transvalvular gradient across aortic valve prosthesis<25 mmHg | Baseline 6 weeks postoperative
  Mild stenosis gradient 25 mmHg, Moderate stenosis gradient 25-40 mmHg, Sever stenosis gradient >40 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed mahmoud ahmed, Doctor, Principal Investigator — Lecturer of cardiothoracic surgery, Faculty of Medicine, Assiut University, Assiut, Egypt

REFERENCES:
- [Background] Dumani S, Likaj E, Dibra L, Llazo S, Refatllari A. Aortic Annular Enlargement during Aortic Valve Replacement. Open Access Maced J Med Sci. 2016 Sep 15;4(3):455-457. doi: 10.3889/oamjms.2016.098. Epub 2016 Sep 2. PMID 27703574
- [Background] Rocha RV, Manlhiot C, Feindel CM, Yau TM, Mueller B, David TE, Ouzounian M. Surgical Enlargement of the Aortic Root Does Not Increase the Operative Risk of Aortic Valve Replacement. Circulation. 2018 Apr 10;137(15):1585-1594. doi: 10.1161/CIRCULATIONAHA.117.030525. Epub 2017 Nov 22. PMID 29167226